CLINICAL TRIAL: NCT05395845
Title: Value of Platelet-Rich Plasma in Post Severe Acute Respiratory Syndrome Coronavirus 2 Smell Disorders
Brief Title: Value of Platelet-Rich Plasma in Post Severe Acute Respiratory Syndrome Coronavirus 2
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aya abdelnasser hassani (Other)
Responsible Party: Sponsor-Investigator, Aya abdelnasser hassani, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP in anosmia
Record Dates: First submitted 2022-03-06; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Anosmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- value of platlet rich plasma (Experimental)
  Interventions: Biological: platelets rich plasma

INTERVENTIONS:
Biological: platelets rich plasma — local ingection of platelets rich plasma

SUMMARY:
The study will be conducted to evaluate :

The efficacy of Platelet Rich plasma in treatment of smell disorders post severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) via the growth factors involved in accelerating and enhancing healing.

DETAILED DESCRIPTION:
Smell is essential sensory function for good quality of life as its preservation helps in identifying several harmful odors .

Viral URTIs can lead to olfactory disorders of varying degree and duration 70% of URTI caused by rhinovirus, adenovirus ,influenza and parainfluanza virus Smell disorders are divided into two types Quantitative (anosmia and hyposmia) Qualitative (parosmia and phantosmia) Anosmia is a total loss of smell . hyposmia is a decrease in the sense of smell. parosmia is a distortion of the smell in presence of an existing stimulus . Phantosmia (Cacosmia) is distortion of the smell in absence of an existing stimulus severe acute respiratory syndrome coronavirus2 (SARS-coV-2)which is a global pandemic started in china 2019 one of respiratory tract infection that affect olfaction and cause varying types of smell impairment.

Smell disorders seem to be more common in SARS-coV2 than other respiratory infections as in some patient persist for long time after resolution of respiratory symptoms Current evidence suggest that olfactory impairment results from propensity of SARS-coV2 for neuroinvasion and neurotrophic activities .

Majority of patients experience some level of smell impairment most often temporary as olfactory neuroepithelium has regenerative power .

European study published on 16 July 2020 reported that some patient affected by SARS -coV2 come solely with olfactory symptoms and most of patient recovered within 2 weeks ,smell not recovered in one quarter of patient 15 Once olfactory dysfunction persists more than 2 weeks a therapy should be considered to avoid persistent impairment of smell One of therapies can be used in ttt of smell disorders ( Platelet _rich plasma) PRP is a process in which a small amount of blood from test subject is separated by special centrifugation process.

PRP contains many growth factor which have a neuroregenerative feature as well as therapeutic effect

ELIGIBILITY:
Inclusion Criteria:

1. patient age above 18 who suffer from anosmia post severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2 more than two weeks
2. Normal airway passage
3. CT Nose and Para nasal sinuses does not show any nasal lesion

Exclusion Criteria:

1. Lesions obstruct airway as nasal polyps, tumors, chronic sinusitis and severe nasal septum deviation
2. Previous Sino nasal surgery
3. Atrophic rhinitis
4. Diabetic patients and those with medical history of bleeding disorders
5. Recieving any medication affect platelets or bone marrow function for 2 weeks prior to testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Loss of Smell on the Olfactory Determination etermination Rating scale for COVID-19 (ODoR-19) at 6 Weeks | baseline
  40 of Participants With Treatment will be improved

REFERENCES:
- [Background] Baig AM, Khaleeq A, Ali U, Syeda H. Evidence of the COVID-19 Virus Targeting the CNS: Tissue Distribution, Host-Virus Interaction, and Proposed Neurotropic Mechanisms. ACS Chem Neurosci. 2020 Apr 1;11(7):995-998. doi: 10.1021/acschemneuro.0c00122. Epub 2020 Mar 13. PMID 32167747
- [Background] Chen X, Fang H, Schwob JE. Multipotency of purified, transplanted globose basal cells in olfactory epithelium. J Comp Neurol. 2004 Feb 16;469(4):457-74. doi: 10.1002/cne.11031. PMID 14755529
- [Background] Woo SH, Jeong HS, Kim JP, Koh EH, Lee SU, Jin SM, Kim DH, Sohn JH, Lee SH. Favorable vocal fold wound healing induced by platelet-rich plasma injection. Clin Exp Otorhinolaryngol. 2014 Mar;7(1):47-52. doi: 10.3342/ceo.2014.7.1.47. Epub 2014 Feb 5. PMID 24587881